CLINICAL TRIAL: NCT03206567
Title: A 6-Month, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Ability and Safety of a Nutraceutical Supplement With Standardized Botanicals to Promote Hair Growth in Women With Self-Perceived Thinning Hair
Brief Title: Efficacy and Safety of a Nutraceutical Supplement With Standardized Botanicals in Women With Thinning Hair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ablon Skin Institute Research Center (Other)
Collaborators: Nutraceutical Wellness Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASIRC-NW-01
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2018-07

CONDITIONS: Hair Thinning
Keywords: Hair thinning, Hair loss, Women, Nutraceutical supplement
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nutrafol Supplement capsules (Active Comparator): Subjects to take four (4) Nutrafol Supplement capsules by mouth daily for 180 days with a substantial meal
  Interventions: Dietary Supplement: Nutrafol Supplement capsules
- Placebo Capsules (Placebo Comparator): Subjects to take four (4) Placebo capsules by mouth daily for 180 days with a substantial meal.
  Interventions: Other: Placebo capsules

INTERVENTIONS:
Dietary Supplement: Nutrafol Supplement capsules — NUTRAFOL's Synergen Complex® is a patent-pending formulation of botanicals with potent anti-inflammatory, anti-stress adaptogenic, antioxidant and DHT-inhibiting properties - combined to synergistically combat the multiple underlying factors that compromise hair growth and health. Some patented ingredients include Sensoril Ashwagandha, BCM-95 BioCurcumin, USPlus Saw Palmetto, EVNolMax 20% Tocotrienol/Tocopherol complex, Bioperine (piperine), Cynatine HNS (solubilized keratin), and Capsimax (capsaicin), all of which are standardized and clinically tested. the Nutrafol supplement capsules are compared to the placebo capsules which contain no active ingredients. Four (4) capsules are taken by mouth once daily with a substantial meal.
  Arms: Nutrafol Supplement capsules
Other: Placebo capsules — The placebo capsules contain no active ingredients. Four (4) capsules are taken by mouth once daily with a substantial meal.
  Arms: Placebo Capsules

SUMMARY:
NUTRAFOL® is a novel nutraceutical supplement, scientifically formulated to specifically target the multiple underlying causes of hair loss and thinning in women. It does not contain hormones, drugs, or industry by-products.

The purpose of this clinical research study is to evaluate the safety, efficacy and physiological effects of NUTRAFOL® supplement compared to placebo in forty (40) female subjects, ages 21-65 years of age with self-perceived thinning hair over the course of six months of continued use.

DETAILED DESCRIPTION:
NUTRAFOL's Synergen Complex® is a patent-pending formulation of botanicals with potent anti-inflammatory, anti-stress adaptogenic, antioxidant and DHT-inhibiting properties - combined to synergistically combat the multiple underlying factors that compromise hair growth and health. Some patented ingredients include Sensoril Ashwagandha, BCM-95 BioCurcumin, USPlus Saw Palmetto, EVNolMax 20% Tocotrienol/Tocopherol complex, Bioperine (piperine), Cynatine HNS (solubilized keratin), and Capsimax (capsaicin), all of which are standardized and clinically tested.

Ingestion of NUTRAFOL® supplement over a six (6) month period will strengthen and promote the growth of hairs in female subjects, ages 21-65 years of age with self-perceived thinning hair when compared to using the placebo tablet. The primary endpoints will be favorable analysis using the Canon Power Shot G16 with 3GEN Dermlite FOTO Pro for macrophotography hair count analysis of terminal and vellus hairs at the three (3) month and six (6) month visits. The secondary endpoints will be favorable improvement in terminal hair diameter measured by the Dino-Lite Digital Microscopic, favorable improvement in the Hair Check device hair bundle measurement for Hair Mass Index (HMI), favorable improvement in the Blinded Physician Global Hair Assessments for hair growth and hair quality, statistically significant positive feedback on the Women's Hair Loss Quality of Life, Self-Assessment and Subject Treatment Satisfaction and Ease of Use questionnaires after six (6) months of NUTRAFOL® supplement or placebo ingestion. See Table of Study Procedures.

All patients enrolled must be identifiable throughout the study. The Investigator will maintain a personal list of patient numbers and patient names to enable records to be found at a later date and the list will be stored in a locked cabinet. Subject numbers consist of a 2 digit number from 01 to 40. Patients will be randomized to active or placebo supplements (2:1 ratio, 26 active and 14 placebo) using a randomization table prepared prior to the start of the study by a non-participating staff member at the office of the Investigator. The study blind will not be broken until the end of the study. All test product and placebo will be labeled with subject numbers per the non-participating staff member. Subjects will be assigned a subject number in numerical order as enrolled. Randomization will occur by assignment to either NUTRAFOL® supplement or placebo with 2:1 ratio (26 active and 14 placebo). Subjects who terminate their study participation for any reason, regardless of whether study medication was used or not, will retain their randomization number.

Visit Procedures: Pre-Study Procedures

1. Candidate subjects will be screened with the eligibility requirements by telephone prior to Visit 1.
2. Candidate subjects will be assigned an appointment time for visiting the clinic.

Visit 1: Baseline, Day 0

1. Individuals will be given an informed consent (IC) document & photographic release form, HIPAA form, confidentiality agreement to read. They will have all of their study related questions answered by the Investigator or his/her designated staff and if they agree, they will sign two copies of the IC/Photography release form, two copies of the HIPAA form, and one copy of the confidentiality agreement. Subjects will be given one copy of the signed IC/Photography release and of the HIPAA agreement to keep, with one copy of each document remaining at the testing facility in the subject's file.
2. Investigator and/or Study Coordinator will review with subject and complete the checklist for all inclusion and exclusion criteria.
3. Investigator and/or Study Coordinator will review with subject and complete the checklist for medical history and concomitant medications.
4. Investigator and/or Study Coordinator will review with subject and complete the General Lifestyle Questionnaire. The General Lifestyle Questionnaire may be found in Appendix VI.
5. Subjects will be given a Women's Hair Loss Quality of Life Questionnaire to read and complete. The Quality of Life Questionnaire may be found in Appendix VII.
6. Candidate subjects will receive a brief physical exam, including examination of the scalp, to rule out any immediately observable medical issues and any scalp alopecias/scalp disorders that are unacceptable for qualification. The physical will additionally include vital signs (pulse and blood pressure), weight and height.
7. Candidate subjects of childbearing potential will complete a urine pregnancy test prior to product distribution.
8. Candidate subjects who have completed all the initial paperwork and meet the inclusion/exclusion qualifications (to include findings of the physical exam) will be assigned a unique subject number. Subjects will be randomized to treatment group prior to dispensing the test product.
9. Qualified subjects will have 2D digital photography of the entire head/hair region for overall general hair growth and fullness (see Appendix I).
10. Qualified subjects will have their scalp prepared for digital macrophotography and initial target area measurements done (see Appendix II).
11. Subjects will have the selected target area (1cm x 1cm) photographed (see Appendix II).
12. Subjects will have the extended target area (2cm x 2cm) bundle of hair measured for Hair Mass Index (HMI) (see Appendix III).
13. Subjects will have ten (10) terminal hairs in a selected test site cut at the base of the scalp and the diameter of the hairs measured (see Appendix IV).
14. Subjects will be dispensed a three (3) month supply of the test product (NUTRAFOL® supplement or Placebo, as randomized) and given written and verbal Usage and Lifestyle instructions (see Appendix X) and a calendar of future visits. Subjects will be instructed to ingest the test product per Sponsor instructions.

Usage Instructions:

Take 4 capsules once daily, along with a meal or immediately following (within 5 minuntes) at approximately the same time of the day, every day. Do not take on an empty stomach. If you forgot to take your dose during a meal, do not skip the dose, take it with something fatty, like peanut butter or coconut oil when you remember. Store at room temperature, in a cool dry location. Do not take if broken or seal is compromised.

Subjects will be instructed to return all empty bottles and unused test product at Visits 2 and 3.

Lifestyle Instructions:

Subjects will be instructed to maintain their normal hair care routine. Subjects will be instructed to use the same brand/type of hair care products and maintain the same haircut, color and style for the study duration.

Subjects who have color treated hair will also be instructed to have the color treatment performed at the same time interval prior to each visit (ie. If on Visit 1, the color treatment was done one week prior then the color treatment is expected to occur at a similar interval of one week prior to Visits 2 and 3).

Subjects will be instructed to come to each visit with clean and dry hair.

Subjects will be instructed to use a medically sound form of birth control during the study.

Visit 2: Month 3 (90 days) ± 1 week (7 days)

1. A clinician will ask subjects if they have experienced any changes in their health or taken new/adjusted current medications since the last visit. If an AE or SAE is reported, the examining Investigator will be informed and the appropriate forms will be completed.
2. The test product will be collected and counted for compliance. Subjects found to be consistently out of compliance will be reminded of the correct usage instructions.
3. Subjects will receive a brief physical exam. The physical will include vital signs (pulse and blood pressure).
4. Subjects will complete the Women's Hair Loss Quality of Life Questionnaire (see Appendix VII), the Self-Assessment Questionnaire (see Appendix VIII) and the Subject Treatment Satisfaction and Ease of Use Questionnaire (see Appendix IX).
5. Subjects will have their hair assessed by the Blinded Investigator for Hair Growth and Hair Quality (see Appendix V).
6. Subjects will have 2D digital photography of the entire head/hair region for overall general hair growth and fullness ( see Appendix I).
7. Subjects will have their scalp prepared for digital macrophotography and target area measurements done (see Appendix II).
8. Subjects will have the selected target area (1cm x 1cm) photographed (see Appendix II).
9. Subjects will have the extended target area (2cm x 2cm) bundle of hair measured for Hair Mass Index (HMI) (see Appendix III).
10. Subjects will have ten (10) terminal hairs in a selected test site cut at the base of the scalp and the diameter of the hairs measured (see Appendix IV).
11. Subjects will be dispensed a three (3) month supply of the test product (NUTRAFOL® supplement or Placebo, as randomized) and given written and verbal Usage and Lifestyle instructions (see Appendix X) and a calendar of future visits. Subjects will be instructed to ingest the test product per Sponsor instructions.

Visit 3: Month 6 (180 days) ± 1 week (7 days)

1. A clinician will ask subjects if they have experienced any changes in their health or taken new/adjusted current medications since the last visit. If an AE or SAE is reported, the examining Investigator will be informed and the appropriate forms will be completed.
2. The test product will be collected and counted.
3. Subjects will receive a brief physical exam. The physical will include vital signs (pulse and blood pressure).
4. Subjects will complete the Women's Hair Loss Quality of Life Questionnaire (see Appendix VII), the Self-Assessment Questionnaire (see Appendix VIII) and the Subject Treatment Satisfaction and Ease of Use Questionnaire (see Appendix IX).
5. Subjects will have their hair assessed by the Blinded Investigator for Hair Growth and Hair Quality (see Appendix V).
6. Subjects will have 2D digital photography of the entire head/hair region for overall general hair growth and fullness (see Appendix I).
7. Subjects will have their scalp prepared for digital macrophotography and target area measurements done (see Appendix II).
8. Subjects will have the selected target area (1cm x 1cm) photographed (see Appendix II).
9. Subjects will have the extended target area (2cm x 2cm) bundle of hair measured for Hair Mass Index (HMI) (see Appendix III).
10. Subjects will have ten (10) terminal hairs in a selected test site cut at the base of the scalp and the diameter of the hairs measured (see Appendix IV).

All primary and secondary parameters will be collected at Visits 1, 2 and 3. Missing data values will be minimized by intensive training of the interviewers in techniques of clarifying answers and checking questionnaires while participants are on-site. When missing values are identified, several approaches such as rescheduled within 24 hours of completion of tests or interviews will be employed to acquire the necessary data. Missing data will be also examined to assess randomness. Descriptive statistics will be obtained for all variables, tests of normality of continuous measures will be made and data will be examined for homogeneity of variance. An appropriate statistical method will be employed to correct for any abnormalities. The comparability of the two treatment groups in baseline demographic and clinical features will be tested with analyses of variance (ANOVAs) for continuous variables and Chi-square analyses for dichotomous variables. Initially, groups will be compared across all three visits for overall interaction effect. For any outcome with significant two-way interaction, group differences from baseline Visit to other two visits will be tested using analyses of variance with repeated measurements. These analyses were performed using the SPSS version 19. All analyses were two-tailed, where applicable, with p-value of 0.05 or less is obtained but other p-values may be evaluated on a case-by-case basis

ELIGIBILITY:
Inclusion Criteria:

1. Females, ages 21-65 years of age.
2. Clinically-determined general good health as determined by responses to the initial study assessment.
3. Females with self-perceived thinning hair as determined on initial study assessment by the Investigator (This will not include patients with medically diagnosed telogen effluvium).
4. Females willing to maintain their normal hair shampooing frequency.
5. Females willing to add the provided oral supplement to their current daily routine.
6. Females willing to not substantially change their current diet, medications, or exercise routines for the duration of the study. If a subject receives physician guidance during the study to change diet, medications, or exercise routine, the subject will need to notify the clinic as soon as possible.
7. Females willing to undergo a brief physical exam to include height, weight, blood pressure, pulse, general physical findings and a scalp exam. The physical exam will occur at Visits 1, 2 and 3.
8. Women of child bearing potential should be willing to have a urine pregnancy test and will comply with a medically sound contraception method (including barrier control, abstinence, etc.). Women who are on birth control should have been on it for at least 6 months and willing to continue the same method of birth control. The initiation of birth control should not have been associated with the initiation of hair loss/thinning.
9. Females with Fitzpatrick I-IV photo skin types.
10. Willingness to have 2D digital photography of the entire head/hair region for overall evaluation of general hair growth and fullness at Visits 1, 2 and 3.
11. Willingness to have digital macrophotography of the target area and scalp for hair counts at Visits 1, 2 and 3.
12. Willingness to have a bundle of hair measured by the Hair Check device for Hair Mass Index (HMI) at Visits 1, 2 and 3.
13. Willingness to have ten (10) terminal hairs from the target area cut at the base of the scalp for microscopic hair measurements at Visits 1, 2 and 3.
14. Willingness to maintain a consistent hair cut and hair color throughout the 6 month study period and to come to visits with clean, dry hair.
15. Willingness of subjects who have color treated hair to have the color treatment performed at the same time interval prior to each visit (ie. If on Visit 1 the color treatment was done one week prior then the color treatment is expected to occur at a similar interval of one week prior to Visits 2 and 3).

Exclusion Criteria:

1. Females with any known allergy or sensitivity to any shampoo/conditioner.
2. Females who are nursing, pregnant, planning to become pregnant during the study.
3. Females with known stressful incident within the last six months (ie. death in family, miscarriage)
4. Females who are participating on any clinical research study at ASIRC or at another research center or doctor's office.
5. Females who have recently (within the last 6 months) started the use of hormones for birth control or hormone replacement therapy (HRT). Women currently using hormones for birth control or HRT must have been on a stable dose (6 months or longer) in order to be eligible for the study (the initiation of HRT or birth control should not have been associated with the initiation of hair loss/thinning).
6. Females currently using any Low Level Laser Therapy (LLLT) to treat thinning hair.
7. Females who have regularly used Rogaine (Minoxidil) within the last 3 months.
8. Females who have used prescription drugs known to affect the hair growth cycle within the last 6 months (e.g., hormone-based birth control for less than 6 months, cyproterone acetate, aldactone/spironolactone, Finasteride or any 5-alpha-reductase inhibitor).
9. Females suffering from other hair loss disorders, such as alopecia areata, scarring alopecia, androgenetic alopecia and telogen effluvium as determined on initial study assessment by the Investigator.
10. No history of burning, flaking, itching, and stinging of the scalp.
11. History of malignancy (except scc and bcc skin cancers) or undergoing chemotherapy or radiation treatments.
12. A known history of autoimmune thyroid disease, any other thyroid disorder/abnormality or other autoimmune disorders that are not controlled in the opinion of the investigator may interfere with the study treatment.
13. A known history of depression or bi-polar disease or any other condition that may impact the subject's participation.
14. Is involved in any injury litigation claims.
15. Known history or recent blood work indicating iron deficiency, bleeding disorders or platelet dysfunction syndrome as well as subjects taking anticoagulant therapy, antiplatelet medications, more than one (1) 325 mg ASA on a daily basis or smokers with usage >20 cigarettes/day.
16. Individuals with self-reported uncontrolled diseases (i.e. diabetes, hypertension, hyperthyroidism, hypothyroidism, etc.). Medical conditions that are under control with or without treatment will be considered on an individual basis by the Investigator.
17. Females with self-reported active hepatitis, immune deficiency, HIV or autoimmune disease.
18. Females having a known active dermatologic condition which, in the opinion of the examining Investigators, might place the subject at a greater risk or interfere with clinical evaluations (e.g., seborrheic dermatitis, psoriasis, atopic dermatitis, advanced skin cancer, etc.).
19. Use of any medications that are known to potentially cause hair loss or affect hair growth, as determined by PI.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2017-12-10 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Number of terminal hairs in the target area of the scalp. | 180 days
  The first primary efficacy parameter from the digital macrophotographs will be the number of terminal hairs in the target area of the scalp. Terminal hair is defined as coarse hair, short or long, found on the scalp with minimum cross-sectional diameter of greater than 40 micrometers. Digital macrophotographs will be taken of the selected target area (1 cm by 1 cm) of each subject at each visit as specified under the Schedule of Procedures. The digital macrophotographs will show the five black colored markings on the scalp that define the target area. Digital macrophotographs will be performed using a Canon Power Shot G16 with 3GEN Dermlite FOTO Pro system.The macrophotographs are then read by the investigator to determine the terminal hair count.
Number of vellus hairs in the target area of the scalp. | 180 days
  The second primary efficacy parameter from the digital macrophotographs will be the number of vellus hairs in the target area of the scalp. Vellus hair is defined as fine, short hairs found on the scalp with maximum cross-sectional diameter of 40 micrometers. Digital macrophotographs will be taken of the selected target area (1 cm by 1 cm) of each subject at each visit as specified under the Schedule of Procedures. The digital macrophotographs will show the five black colored markings on the scalp that define the target area. Digital macrophotographs will be performed using a Canon Power Shot G16 with 3GEN Dermlite FOTO Pro system. The macrophotographs are then read by the investigator to determine the vellus hair count.

SECONDARY OUTCOMES:
Dino-Lite microscopic photographs for terminal hair diameter measurements in the target area. | 180 days
  Dino-Lite Microscopic digital photographs to measure the diameter of the hair will be taken of the selected target area of each subject at each visit as specified under the Schedule of Procedures. Ten (10) terminal hairs just on the border of the 2 cm x 2 cm area used for the Hair Check HMI will be randomly chosen (not all from one direct area) and cut at the surface of the scalp thus not creating any bald patches. The hair diameter will then be measured at 1mm from the cut end of the hair. All calibrations and measurement will be done at the setting of 230X. The ten (10) hair measurements will then be recorded in the source and averaged to attain a median hair diameter for the target area.
Hair Check device hair bundle measurement for Hair Mass Index (HMI). | 180 days
  After attaining the target site (see target site selection section) and the four outer markings this will indicate the target area of 1 cm by 1 cm. Then the Hair Check 4-legged (2 cm x 2 cm) marking template will be placed around the triangulation point and target area. This 2 x 2 cm area will now be used for the creation of the bundle of hair to be measured for Hair Mass Index (HMI).
Quality of Life Questionnaire | 180 days
  Questionnaire about the subjects and how their life is affected by thinning hair.
General Lifestyle Questionnaire | 180 days
  Questionnaire about the subjects general lifestyle and how their life is affected by thinning hair.
Physician Global Hair Assessment | 180 days
  Investigator Hair Growth Global Improvement Scale:
  The treating investigator will complete this live assessment by circling the number on the scale that corresponds to the description that best fits the current global growth improvement at delinated visits as indicated in the schedule of events. The blinded investigator will complete this assessment during the study at Day 90 and Day 180 visits.
  Investigator Hair Quality Global Improvement Scale:
  The treating investigator will complete this live assessment by circling the number on the scale that corresponds to the description that best fits the current hair quality at delinated visits as indicated in the schedule of events. Assessment grading is to be based upon the investigator's appraisal of hair brittleness, dryness, texture, shine, scalp coverage and overall appearance. The blinded investigator will complete this assessment during the study at Day 90 and Day 180 visits.
Self-Assessment Questionnaire | 180 days
  Questionnaire is the evaluation of the growth and qualities related to the subjects hair.

CONTACTS AND LOCATIONS:
Overall Officials: Glynis Ablon, MD, FAAD, Principal Investigator — Ablon Skin Institute Research Center
Locations (1):
- Ablon Skin Institute & Research Center, Manhattan Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ablon G, Kogan S. A Six-Month, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of a Nutraceutical Supplement for Promoting Hair Growth in Women With Self-Perceived Thinning Hair. J Drugs Dermatol. 2018 May 1;17(5):558-565. PMID 29742189